CLINICAL TRIAL: NCT02323282
Title: The Study of Ropivacaine Median Effective Concentration in Ultrasound-guided Supraclavicular Brachial Plexus Block
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yu Shan (Other)
Responsible Party: Sponsor-Investigator, Yu Shan, The study of ropivacaine median effective concentration in ultrasound-guided supraclavicular brachial plexus block, Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Organization: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: Yu Shan
Record Dates: First submitted 2014-10-05; First posted 2014-12-23 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-10

CONDITIONS: Anesthesia
Keywords: Dose-response relationship; Drug
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant

ARMS (1):
- ropivacine (Other)
  Interventions: Drug: ropivacaine

INTERVENTIONS:
Drug: ropivacaine

SUMMARY:
To determine the median effective concentration of ropivacaine hydrochloride for ultrasound-guided supraclavicular brachial plexus block. The result can provide reference for choosing appropriate drug concentration in clinical anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II

Exclusion Criteria:

* upper limb paresthesia
* allergic to local anesthetics
* surgery history of clavicle
* BMI>30kg/m^2

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-10; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
the affection of nerve block | 30 minutes
  The anesthetic efficacy of five nerves, respectively named lateral antebrachial cutaneous nerve, medial cutaneous nerve of the forearm, radial nerve, median nerve, and ulnar nerve was assessed within 30 min after anesthesia. The next concentration of ropivacaine was adjusted according to the response of the previous patient using up-down sequential allocation.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology,Sixth People's Hospital, Shanghai, Shanghai Municipality, China